CLINICAL TRIAL: NCT04233372
Title: Evaluation of (Doravirine / Lamivudine / Tenofovir Disoproxil Fumarate) (Delstrigo®) as a New Strategy for Non-occupational Post Exposure Prophylaxis, a Prospective Open Label Study
Acronym: DORAVIPEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DORAVIPEP; 2019-004140-30 (EudraCT Number)
Record Dates: First submitted 2019-12-20; First posted 2020-01-18 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delstrigo (Experimental)
  Interventions: Drug: Delstrigo

INTERVENTIONS:
Drug: Delstrigo — Doravirine / lamivudine / tenofovir disoproxil fumarate (Delstrigo®) 100 mg doravirine, 300 mg lamivudine,300 mg tenofovir disoproxil fumarate equivalent to 245 mg de tenofovir disoproxil.
  1 covered tablet for day .( will be administered 28 days maximum)

SUMMARY:
Subjects who go to emergency room for possible contact to HIV transmission receive Delstrigo as post exposition prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects attending emergency room due to potential HIV exposition of either sex:
* Aged 18 years or more.
* Who have been exposed to non-occupational HIV and who meet the prerequisites for the current recommendations to begin prophylaxis post-exposition with three antiretroviral drugs.
* Who after being fully informed, give their written consent to participate in the study and undergo the tests and examinations required.
* Individuals able to do follow up correctly.

Exclusion Criteria:

* Pregnant women or nursing mothers or women trying to conceive during the study period.
* Patients in whom it is known or suspected that the source case has a resistance to one of the drugs from the study treatment regimens.
* Treatment with drugs that are contraindicated in the study or products that are in the investigational phase.
* Allergic reactions or intolerance to the compounds of the study treatment regiments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Department and HIV & HCV Clinical Research Unit University Hospital Nantes, Nantes, France
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Inciarte A, Ugarte A, Martinez-Rebollar M, Torres B, Fernandez E, Berrocal L, Laguno M, De la Mora L, De Lazzari E, Callau P, Chivite I, Gonzalez-Cordon A, Solbes E, Rico V, Barrero L, Blanco JL, Martinez E, Ambrosioni J, Mallolas J; DORAVIPEP Study Group. Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate for Nonoccupational HIV-1 Postexposure Prophylaxis: A Prospective Open-Label Trial (DORAVIPEP). Open Forum Infect Dis. 2023 Jul 19;10(8):ofad374. doi: 10.1093/ofid/ofad374. eCollection 2023 Aug. PMID 37539061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1535 subjects received PEP prescriptions between September 2020 and February 2022.
Pre-assignment Details: 406 subjects met PEP criteria and were visited in the emergency department of Hospital Clínic of Barcelona.
  1 subject was a screening failure. 6 subjects were excluded after the initial evalution because they didn't meet the selection criteria and/or had multiple entries.
  399 subjects were included and analized in the study.
Groups:
- Delstrigo: Delstrigo: Doravirine / lamivudine / tenofovir disoproxil fumarate (Delstrigo®) 100 mg doravirine, 300 mg lamivudine, 300 mg tenofovir disoproxil fumarate equivalent to 245 mg de tenofovir disoproxil.
  1 covered tablet for day Treatment will be administered 28 days maximum
Period: Overall Study
Arm/Group | Delstrigo
Started | 399
Completed | 285
Not Completed | 114
Not completed — Lost to Follow-up | 104
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 399 participants were analysed for baseline characteristics
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [27 to 36]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 32
  Male | 364
  Non binary | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  North America | 2
  Latin America | 135
  Europe | 231
  Asia | 7
  Africa | 7
  Unknown | 17
Risk assesment [Count of Participants; unit: Participants]
  Low | 1
  Intermediate | 11
  High | 385
  Unknown | 2
Sexual orientation [Count of Participants; unit: Participants]
  Homosexual | 331
  Heterosexual | 53
  Transexual | 11
  Unknown | 4
Previous PEP [Count of Participants; unit: Participants]
  No | 254
  Yes | 138
  Unknown | 7
Hours from the exposure [Median (Inter-Quartile Range); unit: hours] | 24 [13 to 40]
Abused drugs [Count of Participants; unit: Participants]
  No | 259
  Yes | 111
  Unknown | 29
Sexual exposure [Count of Participants; unit: Participants]
  Anal sex | 361
  Vaginal sex | 53
  Oral sex | 343
  Use of condom | 134
  Broken condom | 128
  Blood contact/exchange | 69
  Semen contact/exchange | 202
Previous sexually transmitted infections [Count of Participants; unit: Participants]
  No | 264
  Yes | 126
  Unknown | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Did Not Complete the 28-day PEP Regimen
Description: Proportion of subjects with treatment completion at day 28. Post exposition prophylaxis (PEP) non-completion is considered in cases:
  1. If the subject dies.
  2. Does not go to visits (loss of follow-up)
  3. Change or suspend the treatment under study for any reason.
  4. Consent withdrawal
Time Frame: 28 days
Population: All participants who received at least one dose of PEP (Intention-To-Treat population).
Measure: Count of Participants; unit: Participants
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Participants | 114

2. Secondary Outcome: Type of Clinical and Laboratory Adverse Events During 28-day PEP With DOR/3TC/TDF
Time Frame: 28 days
Population: 123 is the total number of patients that reported AEs. 183 are the total of AE episodes overall in this 123 participants.
Measure: Count of Units; unit: AEs
Units Other Than Participants: AEs
Arm/Group | Delstrigo
Number analyzed (Participants) | 123
Number analyzed (AEs) | 183
AEs
  Mild | 150
  Moderate | 28
  Severe | 5

3. Secondary Outcome: Assess the Baseline Characteristics Associated to Treatment Non-completion.
Description: Baseline characteristics associated to treatment non-completion were identified using logistic regression model selecting variables in a stepwise fashion.The dependent variable was 'Have discontinuated the 28-days treatment'
Time Frame: 28 days
Population: Odds Ratio (95% confidence interval)
Measure: Number (95% Confidence Interval); unit: Odds Ratio (95% confidence interval)
Groups:
- Delstrigo: Alll patients enrolled in the study
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Odds Ratio (95% confidence interval)
  High risk assessment: number analyzed (Participants) | 397
  High risk assessment | 1.20 [0.32 to 4.52]
  Age (in years) | 0.94 [0.91 to 0.97]
  Sex (male) | 0.42 [0.2 to 0.87]
  Sex (non binary) | 0.57 [0.05 to 6.92]
  Sexual orientation (homosexual): number analyzed (Participants) | 395
  Sexual orientation (homosexual) | 0.98 [0.51 to 1.86]
  Sexual orientation (transexual): number analyzed (Participants) | 395
  Sexual orientation (transexual) | 1.45 [0.37 to 5.68]
  European origin: number analyzed (Participants) | 380
  European origin | 0.86 [0.54 to 1.37]
  Previous STI: number analyzed (Participants) | 383
  Previous STI | 0.98 [0.61 to 1.59]
  Previos PEP: number analyzed (Participants) | 392
  Previos PEP | 0.94 [0.59 to 1.51]

4. Secondary Outcome: Incidence of Clinical and Laboratory Adverse Events During 28-day PEP With DOR/3TC/TDF
Time Frame: 28 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Participants | 123

5. Secondary Outcome: Adherence to cART During 28-day PEP Regimen
Description: Adherence to cART was assessed using the Simplified Medication Adherence Questionnaire (SMAQ) at day 7 and week 4. Non-adherence was defined based on questionnaire responses and pill count.
Time Frame: Day 0 to Day 28 (Week 4)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Participants
  Adherence at day 7: number analyzed (Participants) | 350
  Adherence at day 7 | 336
  Adherence day 28: number analyzed (Participants) | 285
  Adherence day 28 | 281

6. Secondary Outcome: Proportion of Subjects That Maintain Follow-up
Description: Absolute frequency and percentage of individuals who performed month 4 (retention rate).
Time Frame: Month 4
Population: All patients enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Participants | 243

7. Secondary Outcome: Rate of HIV Seroconversion
Description: Number of participants who tested positive for HIV during the 12-week follow-up period after completing post-exposure prophylaxis (PEP) with Delstrigo®.
Time Frame: Day 0 to Day 84
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Delstrigo
Number analyzed (Participants) | 399
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (start of treatment) through Week 12 (approximately 84 days).
Description: The study reported a total of 183 adverse event (AE) episodes among 123 participants.
  Events were categorized by system organ class: gastrointestinal (n = 63), neurological (n = 37), and infections (n = 28).
Arm/Group | Delstrigo
All-Cause Mortality (participants affected / at risk) | 0/399
Serious Adverse Events (participants affected / at risk) | 0/399
Other Adverse Events (participants affected / at risk) | 123/399
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delstrigo (N=399)
Diarrhea, Abdominal pain (Gastrointestinal disorders) | 63 (63)
Neurological (Nervous system disorders) | 37 (37)
Infections (Infections and infestations) | 28 (28)

LIMITATIONS AND CAVEATS:
This was a single-arm, open-label study without a comparator group, which limits the ability to attribute outcomes solely to the intervention. Additionally, the number of participants affected per adverse event category was not specified, restricting detailed safety analysis. Follow-up rates decreased over time, potentially impacting data completeness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04233372/Prot_SAP_000.pdf